CLINICAL TRIAL: NCT01023217
Title: Continuation of Lamivudine Plus Adefovir Versus Switching to Entecavir Plus Adefovir in Adults With Chronic Hepatitis B Who Have Resistant Mutants to Lamivudine and Show Suboptimal Response to Combination of Lamivudine Plus Adefovir
Brief Title: Entecavir Plus Adefovir in Lamivudine-Resistant Chronic Hepatitis B Patients Who Fail Lamivudine Plus Adefovir
Acronym: CAESAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Suk Lim, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-2009-0536
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; lamivudine; adefovir; entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir; adefovir dipivoxil; entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adefovir plus Entecavir (Experimental): Adefovir + Entecavir for 104 weeks
  Interventions: Drug: Adefovir; Drug: Entecavir
- Adefovir plus Lamivudine (Active Comparator): Adefovir + Lamivudine for 52 weeks, and thereafter, Adefovir + Entecavir for 52 more weeks
  Interventions: Drug: Adefovir; Drug: Entecavir; Drug: Lamivudine

INTERVENTIONS:
Drug: Adefovir — Adefovir dipivoxil (Hepsera) 10 mg/day orally for 104 weeks
  Other Names: Adefovir dipivoxil (Hepsera)
Drug: Entecavir — Entecavir 1 mg/day orally
  Other Names: Entecavir (Baraclude)
Drug: Lamivudine — Lamivudine (Zeffix) 100 mg/day orally
  Other Names: Lamivudine (Zeffix)
  Arms: Adefovir plus Lamivudine

SUMMARY:
The presence of persistent inadequate or suboptimal virologic response is a strong risk factor for viral resistance and breakthrough and also for disease progression of chronic hepatitis B, and thus, a change in therapy is required. The combination of entecavir (ETV) and adefovir (ADV) is a promising treatment for patients with lamivudine (LAM)-resistance who show suboptimal response to the combination of LAM and ADV.

In this randomized, open labeled trial,the investigators will compare the efficacy of continuation of ADV plus LAM versus switch to ADV plus ETV in adults with LAM-resistant chronic hepatitis B who shows suboptimal response to the combination treatment of ADV and LAM.

DETAILED DESCRIPTION:
In this randomized, open label, two-arm, single center phase IV trial, the investigators will assess and compare the efficacy and safety of continuation of ADV plus LAM versus switching to ADV plus ETV up to 52-weeks in Korean adults with chronic hepatitis B who have resistant mutants to LAM and show suboptimal response to combination of ADV plus LAM.

All study subjects who complete the initial treatments of 52-weeks will be thereafter treated with the combination of ADV plus ETV for 52 more weeks.

Study period: Nov 2009 - October 2012 Patient enrollment period: November 2009 - December 2010

Study protocol

1. Group A (ADV+LAM group): Adefovir (10 mg/day) + Lamivudine (100 mg/day) for 52 weeks, and thereafter, Adefovir (10 mg/day) + Entecavir (1 mg/day) for 52 more weeks
2. Group B (ADV+ETV group): Adefovir (10 mg/day) + Entecavir (1 mg/day) for 104 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 16 to 75 years of age
2. Compensated liver disease(Child-Pugh class A)
3. HBsAg positive at least 6 months or more
4. HBeAg positive or negative
5. Confirmation of Lamivudine-resistance HBV mutation anytime before the study
6. Patients with suboptimal response (HBV DNA > 2000 IU/mL despite combination of Adefovir [10 mg/day] plus Lamivudine [100 mg/day] for 6 months or more). Serum HBV DNA should be determined by the PCR assay at the local laboratory at screening for this study
7. Patient is ambulatory.
8. Patient is willing and able to comply with the study drug regimen and all other study requirements.
9. The patient is willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patient has a history of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC, such as suspicious foci on imaging studies or elevated serum alpha fetoprotein (AFP) levels. In patients with such findings, HCC should be ruled-out prior to randomizing the patient for the present study.
2. Patient previously received oral antiviral agent other than Lamivudine or Adefovir
3. Patient has received interferon or other immunomodulatory treatment for HBV infection within 12 months before screening for this study.
4. Patient has concomitant other chronic viral infection (HCV or HIV)
5. Patient has evidence of renal insufficiency defined as serum creatinine > 1.5 mg/dL
6. Patient has medical condition that requires use of systemic prednisolone or other immunosuppressive agent (including chemotherapeutic agent)
7. Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years.
8. Patient is pregnant or breastfeeding or willing to be pregnant
9. Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.).
10. A history of treated malignancy (other than hepatocellular carcinoma) is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding three years.
11. Clinical signs of decompensated liver disease as indicated by any one of the following:

    * serum bilirubin > 3 mg/dL
    * prothrombin time > 6 seconds prolonged or INR >1.6
    * serum albumin < 2.8 g/dL
    * History of ascites, variceal hemorrhage, or hepatic encephalopathy
    * Child-Pugh score ≥7

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-suk Lim, M.D.,Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, The Meteropolis of Seoul, South Korea

REFERENCES:
- [Derived] Lim YS, Lee JY, Lee D, Shim JH, Lee HC, Lee YS, Suh DJ. Randomized trial of the virologic response during up to two years of entecavir-adefovir combination therapy in multiple-drug-refractory chronic hepatitis B virus patients. Antimicrob Agents Chemother. 2013 Jul;57(7):3369-74. doi: 10.1128/AAC.00587-13. Epub 2013 May 6. PMID 23650172

RESULTS

PARTICIPANT FLOW:
Groups:
- Adefovir Plus Lamivudine: Adefovir (10 mg/day) + Lamivudine (100 mg/day) for 52 weeks, and thereafter, Adefovir (10 mg/day) + Entecavir (1 mg/day) for 52 more weeks
  Adefovir plus Lamivudine: Adefovir (10 mg/day) + Lamivudine (100 mg/day) for 52 weeks, and thereafter, Adefovir (10 mg/day) + Entecavir (1 mg/day) for 52 more weeks
- Adefovir Plus Entecavir: Adefovir (10 mg/day) + Entecavir (1 mg/day) for 104 weeks
  Adefovir plus Entecavir: Adefovir (10 mg/day) + Entecavir (1 mg/day) for 104 weeks
Period: Overall Study
Arm/Group | Adefovir Plus Lamivudine | Adefovir Plus Entecavir
Started | 45 | 45
Completed | 44 | 45
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Lamivudine-resistant CHB patients who had failed to respond to lamivudine plus adefovir combination therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Adefovir Plus Entecavir | Adefovir Plus Lamivudine | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11) | 49 (11) | 47 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 33 | 34 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 45 | 45 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 45 | 45 | 90
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 45 | 45 | 90
Multiple-Drug-Refractory Chronic Hepatitis B Virus Patients [Number; unit: participants] | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Complete Virologic Response (CVR, Serum HBV DNA Undetectable by PCR or Less Than 60 IU/mL)
Time Frame: at week 52 from randomization
Measure: Number; unit: participants
Arm/Group | Adefovir Plus Entecavir | Adefovir Plus Lamivudine
Number analyzed (Participants) | 45 | 45
participants | 13 | 2

2. Secondary Outcome: Reduction in Serum HBV DNA Levels
Time Frame: at week 52 and at week 104 from randomization
Reporting Status: Not Posted

3. Secondary Outcome: Genotypic Resistance to ADV or ETV
Time Frame: at week 52 and at week 104 from randomization
Reporting Status: Not Posted

4. Secondary Outcome: Normalization of ALT Level
Time Frame: at week 52 and at week 104 from randomization
Reporting Status: Not Posted

5. Secondary Outcome: Complete Virologic Response (CVR, Serum HBV DNA Undetectable by PCR or Less Than 60 IU/mL)
Time Frame: at week 104 from randomization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Adefovir Plus Entecavir | Adefovir Plus Lamivudine
Serious Adverse Events (participants affected / at risk) | 2/45 | 2/45
Other Adverse Events (participants affected / at risk) | 5/45 | 5/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adefovir Plus Entecavir (N=45) | Adefovir Plus Lamivudine (N=45)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid cancer (Endocrine disorders) | 1 (1) | 0 (0)
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
rib fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adefovir Plus Entecavir (N=45) | Adefovir Plus Lamivudine (N=45)
URI (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No